CLINICAL TRIAL: NCT04922424
Title: Mechanisms and Interventions to Address Cardiovascular Risk of Gender-affirming Hormone Therapy in Trans Men
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: not funded
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2000030176
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Hypertension; Hyperlipidemias
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: Baseline testing, then each condition (group) will receive atorvastatin or placebo, followed by washout. Then receive the other condition.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant, PI and RA will not know whether the participant is taking the atorvastatin or placebo. Supervising physician will know.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- atorvastatin (Experimental): We are testing that the lipid sensitive statin, atorvastatin treatment will reduce low density lipoprotein cholesterone, sympathetic nerve activity, increase endothelium-dependent vasodilation and improve autonomic function in trans men, while having little impact on cis women.
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): We are testing that the placebo will have little effect on low density lipoprotein cholesterone, sympathetic nerve activity, endothelium-dependent vasodilation, autonomic function in trans men or cis women.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Atorvastatin — Subjects will ingest placebo or ingest 20 mg atorvastatin for 30 days first. We will include 30 days of washout between treatments to minimize any potential carryover effects.
  Arms: atorvastatin
Other: placebo — Subjects will ingest placebo or ingest 20 mg atorvastatin for 30 days first. We will include 30 days of washout between treatments to minimize any potential
  Arms: Placebo

SUMMARY:
Gender-identity differences are becoming increasingly diagnosed in the US and treatment with gender-affirming hormone therapy (GAHT) is associated with improved mental health outcomes. However, GAHT has been associated with cardiovascular risk in adult transgender patients, although mechanisms and treatments have not been explored. Understanding the cardiovascular effects and exploring the potential of a lipid sensitive statin as a potential treatment is important to optimizing safe treatment strategies for transgender men in mitigating this modifiable risk factor, and designing and implementing effective interventions.

DETAILED DESCRIPTION:
In the US approximately 1.4 million men identify as transgender, a number that is likely to increase with greater recognition of this condition. Gender affirming hormone therapy (GAHT), which attempts to more align the physical appearance with the identified gender, is the primary medical intervention for transgender people and is recognized as medically necessary. GAHT has been associated with increased cardiovascular risk (increased blood pressure, dyslipidemia, and endothelial dysfunction) in transgender men receiving androgens, however little is known about the mechanisms for these changes and few interventions have been proposed. We hypothesize that the altered hormonal milieu is the major driver of increased cardiovascular risk in trans men, and the initiation of testosterone will have effects on lipid profiles, blood pressure and endothelial function. In addition, androgen exposure within the female vascular system is associated with sympathetic nervous system dysregulation. We propose this dysregulation is mediated through rapid dyslipidemia associated with GAHT in trans men receiving androgens. The first aim of this proposal is to test the hypothesis that testosterone treatment in trans men increases sympathetic activation, blood pressure and endothelial dysfunction. Recent studies have demonstrated that vascular endothelial cells are crucial to the pathogenesis of inflammatory disease. Thus, the cholesterol lowering effects of certain statins appear to be mediated, in part, by their action on the endothelium. Important to these studies, HMG-CoA reductase inhibitors (i.e. lipid dependent statins) not only lower LDL-C, but improve both central sympathetic and peripheral microvascular function. Therefore, our second aim is to test the hypothesis that lipid dependent statin therapy will decrease sympathetic activation and improve endothelial function in trans men taking GAHT indicating that the increased sympathetic activity and endothelial dysfunction are mediated by the increased LDL-C with androgens. Trans men undergoing GAHT and cisgender female controls will be examined twice: at baseline, and again following 30 days of treatment with the lipid dependent statin, atorvastatin, in a randomized cross over design. Using microneurography, measures of sympathetic nerve activity (SNA) in response to stressors will be quantified and analyzed within- and between groups and cardiovascular metrics including beat to beat blood pressure and conduit-level endothelial function will be assessed at baseline and with atorvastatin treatment. These novel and innovative studies will illuminate the sympathetic and vascular changes that accompany GAHT, and our atorvastatin intervention will provide insight into the mechanism for these changes as well as provide a method to reduce these risks in trans men undergoing GAHT. This is a critical gap in our knowledge; once these early changes can be identified and quantified, subsequent studies can track these changes over longer trajectories of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Two groups (n=10 each) of subjects will be recruited to complete this study: 1) trans men between 18 and 35 years; 2) cisgender women between 18 and 35 years (Controls). They will have a body mass index (BMI) 18-30 kg·m-2. Our subjects will be matched on BMI and IR, using hemoglobin A1c and Homeostatic Model Assessment of Insulin Resistance technique (HOMA-IR) in order to isolate testosterone effects from other co-morbidities that may impact BP, sympathetic activity or endothelial function. Subjects will have HbA1c of 4-5.9% and a HOMA-IR of 0.5-1.4 to be included in the study. Subjects who smoke, have diabetes, or BP>140/90 will be excluded. Subjects will not be taking medications during the study, including any insulin sensitizing or CV medications.

Exclusion Criteria:

* Subjects with the following histories or conditions will be excluded from the study:

Gynecologic: a. current or past estrogen-dependent neoplasia, b. unexplained vaginal bleeding, c. history of uterine fibroids, d. current pregnancy, e. known or suspected breast or uterine cancer, f. partial or complete hysterectomy.

Cardiac: a. myocardial infarction, ventricular tachycardia or fibrillation, b. angina, c. valvular disease (mitral insufficiency or stenosis, aortic insufficiency or stenosis), d. congestive heart failure, orthopnea, paroxysmal nocturnal dyspnea, e. current arrhythmias, f. prosthetic valves.

Pulmonary: a. current cigarette smokers, or pipe or cigar smokers, b. chronic obstructive pulmonary disease, c. adult asthma, d. dyspnea on exertion, e. current bronchitis, pneumonia, or tuberculosis, f. lung carcinoma, g. pulmonary embolus, h. deep vein thrombosis.

Vascular: a. claudications or history of peripheral vascular disease, b. abdominal or thoracic aortic aneurysm, or repair of same, c. cerebral aneurysm, vascular malformations, d. hypertension, systolic or diastolic, or strong family history of hypertension.

Gastrointestinal: a. GI malignancy, b. hepatitis or other liver disease, current, c. splenomegaly from any cause, d. Cholecystitis, e. current diverticulosis or diverticulitis, inflammatory bowel disease, ulcerative colitis, Crohn's disease, f. previous gastrointestinal surgery.

Infectious Disease: any ongoing intercurrent infection. Hematologic/Oncologic: a. receiving chemotherapy or radiation therapy, b. any metastatic malignancy, c. anemia (hematocrit < 35), d. thrombocytopenia or thrombocytosis, e. neutropenia, f. hematologic malignancy, g. bleeding dyscrasia.

Neurologic: a. history of cerebral vascular accident with any neurologic sequels, b. uncontrolled seizures (e.g., more than 1 seizure/year), c. transient ischemic attacks, d. dementia, e. neurologic conditions producing dyscoordination, peripheral neuropathy, or myopathy.

Endocrine: a. diabetes mellitus, b. any untreated endocrinopathy. Renal: a. chronic renal diseases, b. any history of renal disease or impairment, c. current urinary tract infection.

Musculoskeletal: a. inflammatory arthritis history (e.g., rheumatoid, psoriatic, Reiters), b. any history of pathologic fractures, including vertebral compression fractures.

Pharmacologic: a. any illegal drug use, b. alcohol use greater than an average of 4 oz/day over 30 days, c. coumadin or heparin use.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — trans men, cis women
Enrollment: 0 (Actual)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
flow mediated vasodilation (FMD) | 30 minutes
  FMD measures endothelial function, measured in % change from baseline arterial diameter after release following a short period of occlusion occlusion. The % change in diameter reflects the ability of the vessel to dilate in response to sheer stress induced by the flow following the release of occlusion. This reflects the function of the endothelium, or release of nitric oxide.
Muscle Sympathetic Nerve activity (MSNA) | 2 hours
  measured using microneurography and expressed in bursts/min or bursts/100 heart beats
Cardiovagal baroreflex sensitivity (BRS) | 2 hours
  This is determined as a function of change in R-R interval (from EKG) over systolic blood pressure during rest and regular breathing. Expressed in Units.
Mental Stress Test | 10 minutes
  While measuring sympathetic nervous system activity (SNS) with microneurography, we ask the subject to count backwards from 200 by 7. This increases SNS. Measured in bursts/min or burst/100 heart beats
Voluntary Breath-Hold | 10 minutes
  While measuring sympathetic nervous system activity (SNS) with microneurography, we ask the subject to hold breath as long as possible without straining. The subject does this twice, with a break in between. This increases SNS. Measured in bursts/min or burst/100 heart beats
Systolic Blood Pressure | 2 hours
  SBP, measured in mmHg
Diastolic Blood Pressure | 2 hours
  DBP, measured in mmHg
serum total cholesterol | 5 minutes
  Measured in ng/dl. Elevated total cholesterol can indicate dyslipidemia.
serum low density lipoprotein (LDL)-C | 5 minutes
  Measured in ng/dl. Elevated LDL-C can indicate dyslipidemia
serum high density lipoprotein (HDL-C) | 5 minutes
  Measured in ng/dl. Low HDL-C can indicate dyslipidemia
plasma endothelin-1, (S[ET-1]) | 5 minutes
  endothelial health, increased ET-1 levels in the blood indicate damage to the endothelium

SECONDARY OUTCOMES:
plasma Catecholamines | 5 minutes
  Measure of norepinephrine in pg/ml is a measure of whole body sympathetic nervous system outflow
serum estradiol (S[E2]) | 5 minutes
  estrogen is measured in pg/ml. This should be suppressed in our trans subjects, and low in our cis subjects. In the latter, low estrogen should indicate the early follicular phase of the menstrual cycle.
serum progesterone (S[P4]) | 5 minutes
  progesterone is measured in pg/ml. This should be suppressed in our trans subjects, and low in our cis subjects. In the latter, low progesterone should indicate the early follicular or ovulatory phases of the menstrual cycle.
serum sex hormone binding globulin (P[SHBG]) | 5 minutes
  measured in pg/ml. This provides us with an indication of how much testosterone is free versus bound in the serum, and thus is available for biological function.
serum testosterone | 5 minutes
  measured in pg/ml. This indicates the level of testosterone in our trans men showing they are receiving treatment. It should be high in our trans men and low in our cis women subjects.
plasma creatinine | 5 minutes
  This is a measure of kidney function. Important for blood pressure regulation

CONTACTS AND LOCATIONS:
Overall Officials: Nina Stachenfeld, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States